CLINICAL TRIAL: NCT04950374
Title: Single Center, Open-label, Non-randomized Clinical Trial to Evaluate the Safety and Efficacy of a Moisturizer Body Lotion and the Safety and Perceived Efficacy of a Lip Moisturizer in Adults With Atopic Dermatitis Presenting Dermatological Lesion.
Brief Title: A Clinical Trial to Evaluate the Safety and Efficacy of a Moisturizer Body Lotion and a Lip Moisturizer in Adults of Atopic Dermatitis.
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study halted prematurely, prior to enrollment of first participant due to change on study design.
Sponsor: Johnson & Johnson Consumer Inc. (J&JCI) (Industry)
Responsible Party: Sponsor
Organization: Johnson & Johnson Consumer and Personal Products Worldwide (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: CCSSKA003745; CCSSKA003745 (Other: Johnson & Johnson Consumer Inc.)
Record Dates: First submitted 2021-06-08; First posted 2021-07-06 (Actual); Last update posted 2021-09-08 (Actual); Status verified 2021-09

CONDITIONS: Atopic Dermatitis
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Moisturizer Body Lotion and Lip Moisturizer Regimen (Experimental): All participants will receive and use both products.
  Interventions: Other: Moisturizer Body Lotion; Other: Lip Moisturizer

INTERVENTIONS:
Other: Moisturizer Body Lotion — The body lotion product is a moisturizing formulation intended for topical use on the whole body and face. It will be applied at least twice daily.
Other: Lip Moisturizer — The lip product is a moisturizing formulation intended for topical use on the lips. It will be applied at least twice daily.

SUMMARY:
This study will test the safety and efficacy of 2 moisturizers: a body lotion and a lip moisturizer. For the moisturizer body lotion, the study aims to determine the tolerance of this product by the study population, and its effects on atopic dermatitis condition, skin hydration, skin barrier, skin microbiome and perceived efficacy. For the lip moisturizer, the study aims to determine the tolerance of this product by the same study population and its effects on the perceived efficacy. Participants will receive both products and use them at home for 21 +/- 2 days.

ELIGIBILITY:
Inclusion Criteria:

* Fitzpatrick Skin Type I to VI;
* Subjects with mild to moderate atopic dermatitis according to the SCORAD index (mild global score (up to 24) and moderate global score (between 25 to 50), presenting dermatological lesions at the initial study visit;
* Generally in good health based on medical history reported by the subject;
* Able to read, write, speak and understand Portuguese;
* Person who signed the Consent for Photograph Release and Informed Consent Form;
* Person who agrees to change their leave on body and lip moisturizers to the products of this study, and agrees to use them throughout the test period;
* Intends to complete the study and is willing and able to follow all study instructions.

Exclusion Criteria:

* Subject who attends the Study Site, on the inclusion visit, with leave on moisturizer applied on the instrumental and microbiome evaluation areas;
* Present the need for systemic treatments (as in severe atopic dermatitis cases) such as the use of oral corticosteroids or other types of systemic treatments, as assessed by the Study Physician;
* Perform topical antimicrobial therapies (such as sodium hypochlorite bath or use of topical antibiotics);
* Perform phototherapy;
* Use of antimicrobial / antibacterial / anti germ soaps or other cosmetic and hygiene products;
* Subject who has used other leave on moisturizers in the test areas (body, face and lip), with the exception of investigational products, and/or who has changed their hygiene products during the study;
* Has known allergies or adverse reactions to common topical skincare products;
* Present a skin condition that may influence the outcome of the study (e.g., psoriasis, active skin cancer, etc);
* Present skin lesions (e.g., ulcers, vesicles) or tattoos in the test areas, with the exception of lesions associated with mild or moderate atopic dermatitis;
* Has self-reported Type 1 or Type 2 diabetes or is taking insulin or another anti-diabetic medication;
* Is taking a medication that would mask an Adverse Event (AE) or confound the study results, including:

Immunosuppressive drugs within 2 months before Visit 1; Immunobiological drugs within 2 months before visit 1; Topical anti-inflammatory steroids (corticosteroids) within 15 days before the visit 1; Topical and systemic immunomodulators (such as Tacrolimus and Pimecrolimus) within 15 days before visit 1; Topical and systemic antibiotics 15 days before the visit 1; Non-steroidal anti-inflammatory drugs within 15 days before Visit 1 ; Antihistamines within 2 weeks before Visit 1;

* Is self-reported to be pregnant or planning to become pregnant during the study;
* Has a history of or a concurrent health/other condition/situation which may put the individual at significant risk, confound the study results, or interfere significantly with the individual's participation in the study;
* Participating simultaneously in another study;
* Is an employee/contractor or immediate family member of the PI, Study Site, or Sponsor;
* History of a confirmed Coronavirus disease (COVID-19) in the past 30 days;
* Contact with a person infected with COVID-19 within 14 days prior to inclusion;
* Any international travel within 14 days of inclusion, including members of the same family;
* Subjects with self-reported symptoms in the past 2 weeks: unexplained cough, shortness of breath / difficulty breathing, fatigue, body aches (headaches, muscle aches, stomach pains), conjunctivitis, loss of smell, loss of taste, lack of appetite, nausea, vomiting, diarrhea, palpitations, fever or pain / tightness in the chest; temperature ≥ 38.0 degrees Celsius/100.4 degrees Fahrenheit measured; use of fever reducers within the last 2 days of each onsite visit.

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2021-07-26 (Estimated); Primary Completion 2021-11-26 (Estimated); Study Completion 2021-12-10 (Estimated)

PRIMARY OUTCOMES:
Change from baseline of scores of erythema to 21 ± 2 days | 21 ± 2 days
  At baseline and at 21 ± 2 days, the study physician will evaluate the whole body (including face) and the lips and score the identified erythemas according to the following intensity scale: 0 (absent); 1 (mild); 2 (moderate); 3 (intense).
  This scale will be used to classify this skin reaction on the whole body (including face), and on the lips. The change from baseline will be evaluated to assess skin tolerance of both study products.
Change from baseline of the scores of peeling to 21 ± 2 days | 21 ± 2 days
  At baseline and at 21 ± 2 days, the study physician will evaluate the whole body (including face) and the lips and score the identified peeling according to the following intensity scale: 0 (absent); 1 (mild); 2 (moderate); 3 (intense).
  This scale will be used to classify this skin reaction on the whole body (including face), and on the lips. The change from baseline will be evaluated to assess skin tolerance of both study products.
Change from baseline of the scores of blistering to 21 ± 2 days | 21 ± 2 days
  At baseline and at 21 ± 2 days, the study physician will evaluate the whole body (including face) and the lips and score the identified blistering according to the following intensity scale: 0 (absent); 1 (mild); 2 (moderate); 3 (intense).
  This scale will be used to classify this skin reaction on the whole body (including face), and on the lips. The change from baseline will be evaluated to assess skin tolerance of both study products.
Change from baseline of the scores to edema to 21 ± 2 days | 21 ± 2 days
  At baseline and at 21 ± 2 days, the study physician will evaluate the whole body (including face) and the lips and score the identified edema according to the following intensity scale: 0 (absent); 1 (mild); 2 (moderate); 3 (intense).
  This scale will be used to classify this skin reaction on the whole body (including face), and on the lips. The change from baseline will be evaluated to assess skin tolerance of both study products.
Percentage of participants with Adverse Events through 21 ± 2 days | Up to 21 ± 2 days
  The percentage of participants with AEs, serious adverse events (SAEs), AEs leading to discontinuation and AEs related to skin reactions will be evaluated for skin tolerance up to 21 ± 2 days.
Change from baseline of scores of erythema to 5 ± 1 days | 5 ± 1 days
  At baseline and at 5 ± 1 days, the study physician will evaluate the whole body (including face) and the lips and score the identified erythemas according to the following intensity scale: 0 (absent); 1 (mild); 2 (moderate); 3 (intense).
  This scale will be used to classify this skin reaction on the whole body (including face), and on the lips. The change from baseline will be evaluated to assess skin tolerance of both study products.
Change from baseline of the scores of peeling to 5 ± 1 days | 5 ± 1 days
  At baseline and at 5 ± 1 days, the study physician will evaluate the whole body (including face) and the lips and score the identified peeling according to the following intensity scale: 0 (absent); 1 (mild); 2 (moderate); 3 (intense).
  This scale will be used to classify this skin reaction on the whole body (including face), and on the lips. The change from baseline will be evaluated to assess skin tolerance of both study products.
Change from baseline of the scores of blistering to 5 ± 1 days | 5 ± 1 days
  At baseline and at 5 ± 1 days, the study physician will evaluate the whole body (including face) and the lips and score the identified blistering according to the following intensity scale: 0 (absent); 1 (mild); 2 (moderate); 3 (intense).
  This scale will be used to classify this skin reaction on the whole body (including face), and on the lips. The change from baseline will be evaluated to assess skin tolerance of both study products.
Change from baseline of the scores of edema to 5 ± 1 days | 5 ± 1 days
  At baseline and at 5 ± 1 days, the study physician will evaluate the whole body (including face) and the lips and score the identified edema according to the following intensity scale: 0 (absent); 1 (mild); 2 (moderate); 3 (intense).
  This scale will be used to classify this skin reaction on the whole body (including face), and on the lips. The change from baseline will be evaluated to assess skin tolerance of both study products.

SECONDARY OUTCOMES:
Change from baseline of Atopic Dermatitis severity based on Scoring Atopic Dermatitis Index (SCORAD) to 21 ± 2 days | 21 ± 2 days
  Atopic dermatitis (AD) severity based on SCORAD Index will be reported at baseline and 21 ± 2 days. The tool involves not only medical assessment, but also subjective symptom assessments reported by the subject. The index is divided into the following parts, which receives a numerical score: Extension (ares with AD lesions); Intensity of reactions (erythema, edema, exudation/crusts, abrasions, lichenification and dry skin; and Subjective Symptoms (pruritus and sleep loss). To evaluate these parameters, a scale from 0 to 10 is used. At the end, a global classification of AD is automatically attributed to each subject. Lower global scores means that less severe is the AD condition.
  This assessment will be used to determine the effect of the moisturizer body lotion on AD condition of the study population after a period of use.
Change from baseline to 5 ± 1 days of Atopic Dermatitis severity based on Scoring Atopic Dermatitis Index (SCORAD) | 5 ± 1 days
  Atopic dermatitis (AD) severity based on SCORAD Index will be reported at baseline and 5 ± 1 days. The tool involves not only medical assessment, but also subjective symptom assessments reported by the subject. The index is divided into the following parts, which receives a numerical score: Extension (ares with AD lesions); Intensity of reactions (erythema, edema, exudation/crusts, abrasions, lichenification and dry skin; and Subjective Symptoms (pruritus and sleep loss). To evaluate these parameters, a scale from 0 to 10 is used. At the end, a global classification of AD is automatically attributed to each subject. Lower global scores means that less severe is the AD condition.
  This assessment will be used to determine the effect of the moisturizer body lotion on AD condition of the study population after a period of use.
Change from 5 ± 1 days of Atopic Dermatitis severity based on Scoring Atopic Dermatitis Index (SCORAD) to 21 ± 2 days | 5 ± 1 days to 21 ± 2 days
  Atopic dermatitis (AD) severity based on SCORAD Index will be reported at 5 ± 1 days and 21 ± 2 days. The tool involves not only medical assessment, but also subjective symptom assessments reported by the subject. The index is divided into the following parts, which receives a numerical score: Extension (ares with AD lesions); Intensity of reactions (erythema, edema, exudation/crusts, abrasions, lichenification and dry skin; and Subjective Symptoms (pruritus and sleep loss). To evaluate these parameters, a scale from 0 to 10 is used. At the end, a global classification of AD is automatically attributed to each subject. Lower global scores means that less severe is the AD condition.
  This assessment will be used to determine the effect of the moisturizer body lotion on AD condition of the study population after a period of use.
Mean change from baseline to 21 ± 2 days in skin hydration level of areas with and without AD lesions | 21 ± 2 days
  Skin hydration level of areas with and without AD lesions will be measured with corneometer, a recognized device that determine the water content of stratum corneum. This measure will be used to determine the effect of the moisturizer body lotion on skin hydration of the study population after a period of use.
Mean change from baseline to 5 ± 1 days in skin hydration level of areas with and without AD lesions | 5 ± 1 days
  Skin hydration level of areas with and without AD lesions will be measured with corneometer, a recognized device that determine the water content of stratum corneum. This measure will be used to determine the effect of the moisturizer body lotion on skin hydration of the study population after a period of use.
Mean change from 5 ± 1 days to 21 ± 2 days in skin hydration level of areas with and without AD lesions | 5 ± 1 days to 21 ± 2 days
  Skin hydration level of areas with and without AD lesions will be measured with corneometer, a recognized device that determine the water content of stratum corneum. This measure will be used to determine the effect of the moisturizer body lotion on skin hydration of the study population after a period of use.
Mean change from baseline to 21 ± 2 days in transepidermal water loss (TEWL) to assess skin barrier integrity of areas with and without AD lesions | 21 ± 2 days
  Skin barrier integrity of areas with and without AD lesions will be evaluated using a recognized device that determine the transepidermal water loss. Lower levels of TEWL may be related to a more integrate skin barrier. This measure will be used to determine the effect of the moisturizer body lotion on skin barrier of the study population after a period of use.
Mean change from baseline to 5 ± 1 days in transepidermal water loss (TEWL) to assess skin barrier integrity of areas with and without AD lesions | 5 ± 1 days
  Skin barrier integrity of areas with and without AD lesions will be evaluated using a recognized device that determine the transepidermal water loss. Lower levels of TEWL may be related to a more integrate skin barrier. This measure will be used to determine the effect of the moisturizer body lotion on skin barrier of the study population after a period of use.
Mean change from 5 ± 1 days to 21 ± 2 days in transepidermal water loss (TEWL) to assess skin barrier integrity of areas with and without AD lesions | 5 ± 1 days to 21 ± 2 days
  Skin barrier integrity of areas with and without AD lesions will be evaluated using a recognized device that determine the transepidermal water loss. Lower levels of TEWL may be related to a more integrate skin barrier. This measure will be used to determine the effect of the moisturizer body lotion on skin barrier of the study population after a period of use.
Mean change from baseline to 21 ± 2 days in the Patient-Oriented Eczema Measure (POEM) total score to assess AD severity | 21 ± 2 days
  The POEM is a simple, valid, easily interpreted, and reproducible tool for assessing AD and monitoring aspects of the disease that are important to participants with AD. This tool consists in a questionnaire responded by the participants with questions related to seven AD symptoms (itchy skin, sleep disturbance, bleeding skin, skin weeping/oozing, skin flaking, skin cracking, skin dryness/roughness). Participants must respond each questions specifying how many times per week the symptoms occur using the options: none day; 1 to 2 days; 3 to 4 days; 5 to 6 days; every day. Then each response receives the one of the following scores:
  0 = no days;
  1= 1-2 days; 2 = 3-4 days; 3 = 5-6 days 4= every day. In the end, a total score is calculated by the sum of the 7 items (rating from 0 to 28). Higher scores correlates to a more severe AD condition.
  This measure will be used to determine the effect of the moisturizer body lotion on AD condition of the study population after a period of use.
Mean change from baseline to 7 days in the Patient-Oriented Eczema Measure (POEM) total score to assess AD severity | 7 days
  The POEM is a simple, valid, easily interpreted, and reproducible tool for assessing AD and monitoring aspects of the disease that are important to participants with AD. This tool consists in a questionnaire responded by the participants with questions related to seven AD symptoms (itchy skin, sleep disturbance, bleeding skin, skin weeping/oozing, skin flaking, skin cracking, skin dryness/roughness). Participants must respond each questions specifying how many times per week the symptoms occur using the options: none day; 1 to 2 days; 3 to 4 days; 5 to 6 days; every day. Then each response receives the one of the following scores:
  0 = no days;
  1= 1-2 days; 2 = 3-4 days; 3 = 5-6 days 4= every day. In the end, a total score is calculated by the sum of the 7 items (rating from 0 to 28). Higher scores correlates to a more severe AD condition.
  This measure will be used to determine the effect of the moisturizer body lotion on AD condition of the study population after a period of use.
Mean change from baseline to 14 days in the Patient-Oriented Eczema Measure (POEM) total score to assess AD severity | 14 days
  The POEM is a simple, valid, easily interpreted, and reproducible tool for assessing AD and monitoring aspects of the disease that are important to participants with AD. This tool consists in a questionnaire responded by the participants with questions related to seven AD symptoms (itchy skin, sleep disturbance, bleeding skin, skin weeping/oozing, skin flaking, skin cracking, skin dryness/roughness). Participants must respond each questions specifying how many times per week the symptoms occur using the options: none day; 1 to 2 days; 3 to 4 days; 5 to 6 days; every day. Then each response receives the one of the following scores:
  0 = no days;
  1= 1-2 days; 2 = 3-4 days; 3 = 5-6 days 4= every day. In the end, a total score is calculated by the sum of the 7 items (rating from 0 to 28). Higher scores correlates to a more severe AD condition.
  This measure will be used to determine the effect of the moisturizer body lotion on AD condition of the study population after a period of use.
Perceived Efficacy of the quality of life at baseline | Baseline
  Perceived efficacy related to the quality of life will be subjectively evaluated by the participants through a questionnaire with questions related to the impact of AD in the quality of life. Participants will answer each question using the following qualitative scale: Affected very much; moderately affected; affected a little; did not affected.
  This questionnaire will be used to evaluate the impact of AD in the quality of life before investigational product "Moisturizer body lotion" is used. The responses for each questions will be provided as percentages.
Perceived Efficacy in the quality of life at 7 days | 7 days
  Perceived efficacy related to the quality of life will be subjectively evaluated by the participants through a questionnaire with questions related to the improvement in the quality of life after 7 days of moisturizer body lotion usage. Participants will answer each question using the following qualitative scale: Helped very much; moderately helped; helped a little; did not helped.
  This questionnaire will be used to evaluate the impact of the moisturizer body lotion in the quality of life after periods of use of this product. The responses for each questions will be provided as percentages.
Perceived Efficacy in the quality of life at 14 days | 14 days
  Perceived efficacy related to the quality of life will be subjectively evaluated by the participants through a questionnaire with questions related to the improvement in the quality of life after 14 days of moisturizer body lotion usage. Participants will answer each question using the following qualitative scale: Helped very much; moderately helped; helped a little; did not helped.
  This questionnaire will be used to evaluate the impact of the moisturizer body lotion in the quality of life after periods of use of this product. The responses for each questions will be provided as percentages.
Perceived Efficacy in the quality of life at 21 ± 2 days | 21 ± 2 days
  Perceived efficacy related to the quality of life will be subjectively evaluated by the participants through a questionnaire with questions related to the improvement in the quality of life after 21 ± 2 days of moisturizer body lotion usage. Participants will answer each question using the following qualitative scale: Helped very much; moderately helped; helped a little; did not helped.
  This questionnaire will be used to evaluate the impact of the moisturizer body lotion in the quality of life after periods of use of this product.The responses for each questions will be provided as percentages.
Perceived Efficacy of the moisturizer body lotion at 7 days | 7 days
  Perceived efficacy related to the attributes of moisturizer body lotions will be subjectively evaluated by the participants through a questionnaire using the following qualitative scale: totally agree; agree; neither agree, nor disagree; disagree.
  The responses for each questions will be provided as percentages.
Perceived Efficacy of the moisturizer body lotion at 14 days | 14 days
  Perceived efficacy related to the attributes of moisturizer body lotions will be subjectively evaluated by the participants through a questionnaire using the following qualitative scale: totally agree; agree; neither agree, nor disagree; disagree.
  The responses for each questions will be provided as percentages.
Perceived Efficacy of the moisturizer body lotion at 21 ± 2 days | 21 ± 2 days
  Perceived efficacy related to the attributes of moisturizer body lotions will be subjectively evaluated by the participants through a questionnaire using the following qualitative scale: totally agree; agree; neither agree, nor disagree; disagree.
  The responses for each questions will be provided as percentages.
Perceived Efficacy of the lip moisturizer at 7 days | 7 days
  Perceived efficacy related to the attributes of the lip moisturizer will be subjectively evaluated by the participants through a questionnaire using the following qualitative scale: totally agree; agree; neither agree, nor disagree; disagree. The answer option "Not applicable" can be used.
  The responses for each questions will be provided as percentages.
Perceived Efficacy of the lip moisturizer at 21 ± 2 days | 21 ± 2 days
  Perceived efficacy related to the attributes of the lip moisturizer will be subjectively evaluated by the participants through a questionnaire using the following qualitative scale: totally agree; agree; neither agree, nor disagree; disagree. The answer option "Not applicable" can be used.
  The responses for each questions will be provided as percentages.
Determination of types and quantity of bacteria (skin microbiome) of areas with and without AD lesions at baseline | Baseline
  Skin microbiome is a group of microorganisms, including bacteria, present on the skin surface and plays an important role in AD. To evaluate the type and number of bacteria present on the surface of areas with and without AD lesions, a sample will be collected on this areas using a swab. The evaluation will be done through metagenomics, a technique that allows the determination of the types and quantity of bacteria present in an specific area.
  This assessment will be used to determine the effect of the moisturizer body lotion on skin microbiome after a period of use.
Determination of types and quantity of bacteria (skin microbiome) of areas with and without AD lesions at 21 ± 2 days | 21 ± 2 days
  Skin microbiome is a group of microorganisms, including bacteria, present on the skin surface and plays an important role in AD. To evaluate the type and number of bacteria present on the surface of areas with and without AD lesions, a sample will be collected on this areas using a swab. The evaluation will be done through metagenomics, a technique that allows the determination of the types and quantity of bacteria present in an specific area.
  This assessment will be used to determine the effect of the moisturizer body lotion on skin microbiome after a period of use.
Visual skin condition of areas with and without AD lesions at baseline captured photographically | Baseline
  Images of areas with and without AD lesions will be captured through a professional camera at baseline to visualize the skin condition of these areas before the use of moisturizer body lotion.
  No analysis is planned. These images will be used as a qualitative complement to the other results for moisturizer body lotion.
Visual skin condition of areas with and without AD lesions at 5 ± 1 days captured photographically | 5 ± 1 days
  Images of areas with and without AD lesions will be captured through a professional camera at 5 ± 1 days to visualize the skin condition of these areas after the use of moisturizer body lotion.
  No analysis is planned. These images will be used as a qualitative complement to the other results for moisturizer body lotion.
Visual skin condition of areas with and without AD lesions at 21 ± 2 days captured photographically | 21 ± 2 days
  Images of areas with and without AD lesions will be captured through a professional camera at 21 ± 2 days to visualize the skin condition of these areas after the use of moisturizer body lotion.
  No analysis is planned. These images will be used as a qualitative complement to the other results for moisturizer body lotion.
Testimonial regarding the experience with moisturizer body lotion at 21 ± 2 days | 21 ± 2 days
  A testimonial regarding the experience with moisturizer body lotion will be provided by the participants through an open question at the end of the study. The purpose is to know their opinion and experience using this product during the study.

CONTACTS AND LOCATIONS:
Overall Officials: Mariane M Mosca, Bsc, Principal Investigator — Allergisa Pesquisa Dermato-Cosmetica LTDA

IPD SHARING:
Plan to Share IPD: Yes
Johnson & Johnson Consumer Inc. has an agreement with the Yale Open Data Access (YODA) Project to serve as the independent review panel for evaluation of requests for clinical study reports and participant level data from investigators and physicians for scientific research that will advance medical knowledge and public health. Requests for access to the study data can be submitted through the YODA Project site at http://yoda.yale.edu.
URL: http://yoda.yale.edu

REFERENCES:
- [Background] Aoki V, Lorenzini D, Orfali RL, Zaniboni MC, Oliveira ZNP, Rivitti-Machado MC, Takaoka R, Weber MB, Cestari T, Gontijo B, Ramos AMC, Silva CMR, Cestari SDCP, Souto-Mayor S, Carneiro FR, Cerqueira AMM, Laczynski C, Pires MC. Consensus on the therapeutic management of atopic dermatitis - Brazilian Society of Dermatology. An Bras Dermatol. 2019 Apr;94(2 Suppl 1):67-75. doi: 10.1590/abd1806-4841.2019940210. Epub 2019 Jun 3. PMID 31166406
- [Background] Grice EA, Kong HH, Conlan S, Deming CB, Davis J, Young AC; NISC Comparative Sequencing Program; Bouffard GG, Blakesley RW, Murray PR, Green ED, Turner ML, Segre JA. Topographical and temporal diversity of the human skin microbiome. Science. 2009 May 29;324(5931):1190-2. doi: 10.1126/science.1171700. PMID 19478181
- [Background] Gallo RL, Nakatsuji T. Microbial symbiosis with the innate immune defense system of the skin. J Invest Dermatol. 2011 Oct;131(10):1974-80. doi: 10.1038/jid.2011.182. Epub 2011 Jun 23. PMID 21697881
- [Background] Stamatas GN, Capone K. New findings, and the impact of infant skin microbiota on product development. Cosmetics and Toiletries.
- [Background] Brazil. Conselho Nacional da Saúde. Resolution Nº 466, December 2012.
- [Background] Pan-American Health Organization. Good Clinical Practices: American Document. IV Pan-Americana Conference for Harmonization of Pharmaceutical Regulation, 2005.
- [Background] Blichmann CW, Serup J. Assessment of skin moisture. Measurement of electrical conductance, capacitance and transepidermal water loss. Acta Derm Venereol. 1988;68(4):284-90. PMID 2459872
- [Background] Agner T, Serup J. Comparison of two electrical methods for measurement of skin hydration. An experimental study on an irritant patch test reaction.
- [Background] Brazil. Agência Nacional de Vigilância Sanitária (ANVISA). Guideline for Safety Assessment of Cosmetic Products. 2 edition, 2012.
- [Background] Brazil. Agência Nacional de Vigilância Sanitária (ANVISA). Resolution - RDC Nº 10, 03 March 2015.